CLINICAL TRIAL: NCT00957918
Title: Randomized, Double-Blind, Parallel Group, Placebo Controlled Safety, Tolerability and Efficacy Study of NP002 in Subjects With Idiopathic Parkinson's Disease With Dyskinesias Due to Levodopa Therapy
Brief Title: Study of NP002 in Subjects With Idiopathic Parkinson's Disease to Treat Dyskinesias Due to Levodopa Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neuraltus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP002-09-001
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-09

CONDITIONS: Parkinson's Disease
Keywords: levodopa-induced dyskinesia; Parkinson's disease; parkinsonian; levodopa-induced dyskinesias in Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine (Experimental): Active drug is nicotine dihydrate bitartrate, provided as an oral capsule at escalating doses, 1 mg to 6 mg, once every 6 hours
  Interventions: Drug: nicotine
- placebo (Placebo Comparator): Subjects in this arm receive placebo capsules orally
  Interventions: Other: placebo comparator

INTERVENTIONS:
Drug: nicotine — Oral capsule self administered in escalating doses from 1 mg to 6 mg, 4 times a day. Each dose is is taken for two weeks, except the highest dose, which is taken for 4 weeks. At the end of 10 weeks, the dose is tapered down over 9 days. Subject is continued on study through week 14.
  Other Names: NP002
  Arms: Nicotine
Other: placebo comparator — oral capsules containing only excipient will be self-administered with the same regimen as the active drug, 4 times a day, approximately every 6 hours for 10 weeks and nine days. Study is continued through week 14.
  Arms: placebo

SUMMARY:
The study is designed to answer the question: will nicotine at doses that do not cause serious side effects, show feasibility in treatment of levodopa-induced dyskinesia in patients with Parkinson's disease?

DETAILED DESCRIPTION:
Nicotine will be employed at daily doses lower than those available OTC as smoking-cessation patches, in parkinsonian patients experiencing disabling dyskinesias due to their levodopa treatment. The principal adverse effect from this dose level of nicotine is expected to be nausea on acute administration to nicotine-naive patients. Because tolerance to the effects of nicotine is achieved by repeated dose, the study is designed to gradually escalate from 6 to 24 mg per day, taken in 6 separate oral doses of 6 mg each. The study is designed to see if doses which can be tolerated by parkinsonian patients will also reduce the severity and frequency of the dyskinesias experienced following administration of levodopa, the gold standard medication for Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of probable idiopathic Parkinson's disease
* in stable health
* male and female aged 30-83 yrs
* Hoehn and Yahr stage II through IV inclusive
* levodopa-induced dyskinesias present greater than 25% of waking day; rating equal or greater than 2 on item 32 of UPDRS
* dyskinesias moderately or severely disabling as determined by a rating of equal or greater than 2 on item 33 of UPDRS
* Mini-Mental state (MMSE) score of equal or greater than 26
* on a stable dose of levodopa for at least 30 days
* if subjects are taking dopamine antagonists, amantadine, MAO-B inhibitors (rasagiline only) or COMT inhibitors, doses must have been stable for at least 30 days

Exclusion Criteria:

* Secondary or non-idiopathic Parkinson's disease
* Subjects with parkinsonian symptoms who do not respond to levodopa therapy
* history of schizophrenia, or other DSM-IV TR axis 1 diagnosis sufficient to interfere with or affect study conduct or interpretation of results
* any history (past 5 years) of suicide or suicide attempt or thoughts or urges of suicide on direct questioning
* subjects who score 2 or higher on a single module of the Jay MIDI scale
* moderate or severe hallucinations, psychoses or delusions
* any medical condition or lab abnormality presenting an unwarranted risk in the opinion of the Investigator
* history of HIV positivity, AIDS, or active hepatitis determined by subject report
* female who is pregnant or breastfeeding
* female of childbearing potential not using double barrier method of birth control throughout the duration of the study
* receipt of a neurosurgical intervention (e.g. brain surgery)related to Parkinson's disease or any neurosurgical procedure sufficient to interfere with study conduct or interpretation of results
* must not have systolic blood pressure ≥150; diastolic ≥95.
* must not have ECG at screening judged clinically significantly abnormal by investigator
* must not have QTc > 450 msec at ECG screen
* must not have current angina pectoris, history of ventricular arrhythmias, uncontrolled hyperthyroidism, known or suspected pheochromocytoma, symptomatic vasospastic disease, or active peptic ulcer
* must not have a history of stroke, transient ischemic attack (TIA) or myocardial infarction within the last 2 years
* must not have current drug or alcohol abuse within the last two years. Acceptable alcohol use is no more than 3 ounces of alcohol, 3 beers or 2 glasses of wine per day.
* must not be participating in another drug trial or have participated in another drug study in the last 30 days. Observational trials with no intervention are acceptable provided permission is obtained from the other study sponsor in writing.
* must not be unwilling or unable to swallow capsules
* must not have a positive urine test for cotinine at screening
* must not be a smoker, previous (less than 5 years since cessation) smoker or have regular exposure to second hand smoke
* must not be allergic to capsule excipients
* must not be allergic to ondansetron. If allergic, they may participate provided they understand there is no rescue medication for potential nausea or vomiting during the study
* must not have known sensitivity to nicotine or nicotine-containing products
* must not be taking any of the following medications or substances within a minimum of 30 days: nicotine, any form; CYP2A6 inducers or inhibitors during the course of the study or within 30 days of the planned initial dose (your investigator will have a full list of these drugs); Monoamine oxidase inhibitors (with the exception of rasagiline, which is allowed)(your investigator will have a full list of these drugs); apokyn (apomorphine), due to its contraindication with ondansetron); warfarin.

Ages: 30 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
frequency and severity of adverse events, active vs placebo | Every two weeks during dosing (week 0 to week 12) and weekly thereafter for 2 weeks following cessation of dosing
measure of impulse control (rMIDI), active vs placebo | at screening and 4 weeks, 10 weeks, 12 weeks and 14 weeks

SECONDARY OUTCOMES:
measure of frequency and severity of dyskinesia (USDysRS), active vs placebo | At screen and every two weeks through week 10
Parkinson's disease severity (UPDRS part II,III,IV), active vs placebo | At screen and every two weeks through week 10

CONTACTS AND LOCATIONS:
Overall Officials: Abrahan N Lieberman, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Barrow Neurology Clinics
Locations (12):
- United States (12):
  - Barrow Neurology Clinics at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Keck/USC School of Medicine -Department of Neurology, Los Angelis, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Parkinson's Disease & Movement Disorders Ctr of Boca Raton, Boca Raton, Florida
  - Collier Neurologic Specialists, LLC, Naples, Florida
  - Strurers Parkinson's Center, Golden Valley, Minnesota
  - David L. Kreitzman, M.D., P.C., Commack, New York
  - 108-14 72nd Ave, Second floor, Forest Hills, New York
  - Duke University Medical Center, Department of Neurology, Durham, North Carolina
  - The Movement Disordedr Clinic of Oklahoma, Tusla, Oklahoma
  - Parkinson's Disease and Movement Center, Penn Comprehensive Neuroscience Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lieberman A, Lockhart TE, Olson MC, Smith Hussain VA, Frames CW, Sadreddin A, McCauley M, Ludington E. Nicotine Bitartrate Reduces Falls and Freezing of Gait in Parkinson Disease: A Reanalysis. Front Neurol. 2019 May 7;10:424. doi: 10.3389/fneur.2019.00424. eCollection 2019. PMID 31133957